CLINICAL TRIAL: NCT03402516
Title: Impact of the Diameter on the Performance of Two Bipolar Resectors 18.5Fr and 26Fr
Brief Title: Comparison of Two Bipolar Resector in Less Than 3cm Myoma Resection
Acronym: DIAPER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Capmas Perrine, Principal investigator, Bicetre Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-A01740-51
Record Dates: First submitted 2017-12-26; First posted 2018-01-18 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Rate of Complete Resection in a Unique Surgical Time
Keywords: hysteroscopic myomectomy; 26Fr resector; 18.5Fr resector

STUDY DESIGN:
Intervention Model Description: Randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 18.5Fr resector (Experimental): Used of a 18.5Fr bipolar resector for hysteroscopic myomectomy. Cervical dilatation would be performed until Hegar bougie number 7 and then a classic hysteroscopic resection will be performed with a 18.5Fr bipolar resector.
  Interventions: Device: 18.5 resector
- 26Fr resector (Active Comparator): Used of a 26Fr bipolar resector for hysteroscopic myomectomy. Cervical dilatation would be performed until Hegar bougie number 10 and then a classic hysteroscopic resection will be performed with a 24Fr bipolar resector.
  Interventions: Device: 26Fr resector

INTERVENTIONS:
Device: 18.5 resector — hysteroscopic myomectomy with a 18.5 Fr resector after cervical dilatation until Hegar bougie number 7
  Arms: 18.5Fr resector
Device: 26Fr resector — hysteroscopic myomectomy with a 26Fr resector after cervical dilatation until Hegar bougie number 10
  Arms: 26Fr resector

SUMMARY:
Hysteroscopic resection of type 0, 1 or 2 myoma is frequent. The more frequent resector used for myoma resection is 26Fr hysteroscope. Actual miniaturization of resector led to 18.5Fr resector with a potential benefit because of less dilatation. These resectors are often used but no scientific evaluation has been performed.

Hypothesis of this non inferiority trial is that complete resection in a unique surgical time will be comparable with both resectors.

DETAILED DESCRIPTION:
Myoma type 0, 1 or 2 are often symptomatic (abnormal uterine bleeding or infertility) and hysteroscopic resections are thus frequent. This management is a minimally invasive surgery.

Usually, a 26Fr resectoscope is used and the main articles on this topic report hysteroscopie resections with a 26Fr resectoscope. Miniaturization of resector led to decrease in the size of resectors with a potential benefit because of a less important cervical dilatation and then a smaller risk of adverse events and an increase in the number of surgery under local anaesthesia.

Use of 18.5Fr resectors is more and more frequent but, to our knowledge, it has never been evaluated for benefit on cervical dilatation but also for rate of complete resection in one time, surgical length and rate of unbalanced input/output.

Intuitively, a smaller diameter could led to a less traumatic cervical dilatation but it could also led to an higher risk of incomplete treatment in one time and a longer surgical duration and a more frequent unbalanced input/output.

No study compare use of these two resectors (18.5 and 26Fr) all the more randomized. With 26Fr resector, the rate of complete resection in one time for less than 3cm myoma is around 90%. If this rate is higher with the 18.5Fr resector, the risk/benefit balance (including economic evaluation) won't be favorable to this use.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* With a type 0,1 or 2 unique myoma requiring surgery

Exclusion Criteria:

* No medical care

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Comparison with chi square test of rate of complete surgery in one time | 3 years
  Complete resection of myoma in one time

SECONDARY OUTCOMES:
Duration of surgery | 3 years
  Comparison of duration of surgery between 2 arms
Rate of unbalanced in and out balance | 3 years
  Comparison of rate of unbalanced in and out balance between the 2 groups. A in/out balance higher than 500cc will be consider has unbalanced).
Cost effectiveness analyses | 3 years
  Comparison of cost for complete resection of myoma between groups
Complications rate | 3 years
  Comparison of complications rate (including cervical complications)
Use of a 26Fr resector | 3 years
  Report of the rate of use of a 26Fr resector in the 18.5Fr group

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Bicetre, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: Undecided